CLINICAL TRIAL: NCT02699879
Title: Post-Authorisation Safety Study of Esbriet® (Pirfenidone): A Prospective Observational Registry to Evaluate Long-Term Safety in a Real-World Setting
Brief Title: Evaluation of Long-Term Safety of Pirfenidone (Esbriet) in Participants With Idiopathic Pulmonary Fibrosis (IPF)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: WB29908; PIPF-025 (Other: InterMune)
Record Dates: First submitted 2016-02-26; First posted 2016-03-04 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — pirfenidone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Pirfenidone: Participants will receive pirfenidone orally according to the physician discretion.
  Interventions: Drug: Pirfenidone

INTERVENTIONS:
Drug: Pirfenidone — Pirfenidone will be administered according to the physician discretion as part of standard care.
  Other Names: Esbriet

SUMMARY:
This single arm, post-authorisation study is designed to evaluate the long-term safety of pirfenidone in participants with IPF. The enrolment of participants will be completed within approximately 24 months. Participants will receive pirfenidone according to the physician discretion and will be followed for 2 years. Treating physicians will collect pre-specified data at the baseline and every 3 months thereafter, for the duration of the participants' participation in study.

ELIGIBILITY:
Inclusion Criteria:

* A clinical decision has been made, prior to study enrolment, to prescribe Esbriet
* Participants who are newly prescribed Esbriet therapy
* Initiation of Esbriet therapy is not more than 30 days prior to study enrolment

Exclusion Criteria:

* Participants receiving an investigational agent defined as any drug that has not been approved for marketing for any indication in the country of the participating site
* Participant has received Esbriet therapy 30 days or more prior to current treatment course (e.g., prior participation in clinical trials)
* Participant has any contraindication for the use of Esbriet, according to the current local version of the Summary of Product Characteristics (SPC)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants receiving treatment for IPF with pirfenidone according to the physician's discretion
Sampling Method: Non-Probability Sample
Enrollment: 1009 (Actual)
Dates: Start 2012-02-16 (Actual); Primary Completion 2016-09-15 (Actual); Study Completion 2016-09-15 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with clinically significant ADRs of special interest | up to 2 years
Percentage of participants with adverse drug reactions (ADRs) and serious adverse drug reactions | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (106):
- Austria (5):
  - Medical University Graz; Department for Respiratory Diseases, Graz
  - LKH Hohenems; Abteilung für Pulmologie, Hohenems
  - Medizinische Universitat Innsbruck; Department of Internal Medicine, Pneumology Centre, Innsbruck
  - Klinikum Klagenfurt; Abteilung für Pulmologie, Klagenfurt
  - St. Johanns-Spital; Abt. Für Lungenkrankungen, Salzburg
- Denmark (3):
  - Aarhus University Hospital; Lungemed afd. B, Aarhus
  - Gentofte Hospital, Lungemedicinsk Afdeling, Hellerup
  - Odense Universitetshospital, Lungemedicinsk Afdeling J, Odense
- Finland (4):
  - Helsinki University Central Hospital; Dep. of Pulmonary Medicine, Helsinki
  - Kuopio University Hospital, Kuopio
  - Tampere University Hospital; Lung Clinic, Tampere
  - Turku University Hospital; Dept of Pulmonology, Turku
- France (23):
  - CHU Angers,Service de Pneumologie, Angers
  - Hopital Jean Minjoz; Pneumologie, Besançon
  - Hopital Avicenne; Pneumologie, Bobigny
  - Hopital de La Cavale Blanche; Service de Medecine Interne & de Pneumologie, Brest
  - Hopital Louis Pradel; Pneumologie, Bron
  - Hopital Cote De Nacre; Pneumologie, Caen
  - Chu Site Du Bocage;Pneumologie, Dijon
  - CHU de Grenoble; Medecine Aigue Spec, Grenoble
  - Hopital Calmette; Pneumologie, Lille
  - CHU de Limoges, Limoges
  - Hopital Nord AP-HM, Marseille
  - Hopital Nord; Pneumologie, Marseille
  - CHU Montpellier, Montpellier
  - Hopital Saint Louis, Paris
  - Hopital Bichat Claude Bernard ; Service de Pneumologie, Paris
  - HEGP; Pneumologie, Paris
  - Hopital Tenon;Pneumologie, Paris
  - Hôpital Haut-Lévêque - CHU de Bordeaux - Groupe Hospitalier Sud, Pessac
  - Hopital De La Maison Blanche;Maladies Respiratoires, Reims
  - Hopital de Pontchaillou; Service de Pneumologie, Rennes
  - Chu De Strasbourg; Hopital Civil, Strasbourg
  - Hopital Larrey; Pneumologie, Toulouse
  - Chu De Tours,Service de Pneumologie, Tours
- Germany (40):
  - Zentralklinik Bad Berka GmbH; Pneumologie, Bad Berka
  - Lungenklinik Ballenstedt/Harz gGmbH Lungenklinik Ballenstedt/Harz gGmbH, Ballenstedt
  - Evang. Lungenklinik Berlin Klinik für Pneumologie, Berlin
  - Charite - Universitätsmedizin Berlin; Campus Virchow-Klinikum, Med. Klinik m. S. Infekt und Pneumo, Berlin
  - Gemeinschaftskrankenhaus Havelhöhe Klinik f.Innere Medizin Kardiologie Pneumologie, Berlin
  - HELIOS Klinikum Emil von Behring Klinik f.Pneumologie Onkologie u.Infektiologie, Berlin
  - Berufsgenossenschaftliches Uni-Klinikum Bergmannsheil GmbH, Bochum
  - Klinkum Coburg GmbH, Coburg
  - Fachkrankenhaus Coswig GmbH Zentrum f.Pneumologie Beatmungsmedizin Thorax-u.Gefäßchirurgie, Coswig
  - Carl-Thiem-Klinik Cottbus; Medizinische Klinik, Cottbus
  - Klinik Donaustauf Zentrum für Pneumologie, Donaustauf
  - Ruhrlandklinik Lungenzentrum der UNI Essen Abt.Pneumologie-Allergologie, Essen
  - Klinikum Esslingen; Klinik für Kardiologie, Angiologie und Pneumologie, Esslingen am Neckar
  - Klinik Maingau, Frankfurt
  - Studienzentrum/Praxis Dr. Keller Frankfurt, Frankfurt
  - IFS - Interdisziplinäres Facharztzentrum; Institut für klinische Forschung Pneumologie, Frankfurt am Main
  - Universitätsklinikum Freiburg, Abteilung Pneumologie, Freiburg im Breisgau
  - Klinik Schillerhöhe Zentrum f.Pneumologie u.Thoraxchirurgie, Gerlingen
  - Universitätsklinikum Standort Gießen Medizinische Klinik II u. Poliklinik Innere Med./Pneumologie, Giessen
  - Universitätsmedizin Greifswald Klinik für Innere Medizin B und Poliklinik, Greifswald
  - LungenClinic Grosshansdorf GmbH; Zentrum fur Pneumologie und Thoraxchirurgie, Großhansdorf
  - Medizinische Hochschule Hannover, Hanover
  - KRH Klinikum Oststadt-Heidehaus; Pneumologie, Intensiv- und Schlafmedizin, Hanover
  - Lungenklinik Hemer; Abt. Pneumologie, Hemer
  - Universitaetsklinikum des Saarlandes; Innere Medizin V, Homburg/Saar
  - Fachklinik für Lungenerkrankungen, Immenhausen
  - Universitätsklinikum Jena; Medizinische Klinik I, Jena
  - Universitaetsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Universität Leipzig; Medizinische Klinik und Poliklinik I, Abteilung Pneumologie, Leipzig
  - Lungenklinik Lostau gGmbH; Klinik für Pneumologie II, Lostau
  - Klinik Löwenstein gGmbH Medizinische Klinik II, Löwenstein
  - Universitätsklinikum Magdeburg Klinik für Kardiologie Angiologie u.Pneumologie, Magdeburg
  - Klinikum der Universität München; Campus Großhadern; Med. Klinik und Poliklinik V, München
  - Klinikum Nuernberg Nord; Medizinische Klinik 3, Schwerpunkt Pneumologie, Allergologie, Schlafmedizin, Nuremberg
  - RoMed Klinikum Rosenheim, Medizinische Klinik III, Rosenheim
  - Krankenhaus Bethanien gGmbH, Solingen
  - Krankenhaus vom Roten Kreutz; Klinik fuer Pneumologie, Stuttgart
  - Johanniter-Krankenhaus im Fläming Treuenbrietzen GmbH; Fachklinik Pneumologie/ Thoraxchirurgie, Treuenbrietzen
  - Fachkliniken Wangen Medizinische Klinik, Wangen
  - Universitätsklinikum Würzburg, Kinderklinik u. Poliklinik, Würzburg
- Ireland (4):
  - Cork University Hospital, Cork
  - Mater Misecordiae University Hospital, Dublin
  - St Vincents University Hospital, Dublin
  - Galway University Hospital; Department of Respiratory Medicine, Galway
- Italy (7):
  - Ospedale Morgagni-Pierantoni; U.O. Pneumologia, Forlì, Emilia-Romagna
  - A.O. Universitaria Policlinico Di Modena; DIP. Malattie Dell'apparato Respiratorio, Modena, Emilia-Romagna
  - Universita' Degli Studi Di Milano Bicocca, Ospedale Vecchio; facolta di medicina e chirurgia, dipart, Monza, Lombardy
  - A.O. Universitaria San Luigi Gonzaga di Orbassano; Ambulatorio per le Malattie Rare del Polmone, Orbassano (TO), Piedmont
  - Azienda Ospedaliero Universitaria Di Sassari; Clinica Pneumologica, Sassari, Sardinia
  - Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
  - A.O. Univ. Senese Policlinico S. Maria alle Scotte; UOC Malattie Resepiratorie e Trapianto Polmonare, Siena, Tuscany
- Norway (3):
  - Haukeland Hospital - University Of Bergen: Department of Resp Med, Bergen
  - Oslo University Hospital Rikshospitalet; Lungeavdelingen, Oslo
  - St. Olav's Hospital; Lung Clinic, Trondheim
- Sweden (2):
  - Karolinska Universitetssjukhuset Solna; Lung Allergikliniken, Stokholm, Solna
  - Akademiska Sjukhuset; Lungmedicinska Kliniken, Uppsala
- United Kingdom (15):
  - Southmead Hospital; Respiratory Department, Bristol
  - Papworth Hospital NHS Foundation Trust; Respiratory Department, Cambridge
  - Castle Hill Hospital; Respiratory Medicine, Cottingham
  - Royal Devon and Exeter Hospital (Wonford), Exeter
  - Southampton General Hospital; Respiratory Department, Hampshire
  - Glenfield Hospital, Leicester
  - University Hospital Aintree; Pulmonary Vascular Diseases Unit, Liecester
  - University College London Hospital; Respiratory Medicine, London
  - Royal Brompton Hospital; Respiratory Department, London
  - St. Mary'S Hospital; Dept of Medicine, London
  - Wythenshawe Hospital, Manchester
  - Nottingham University Hospitals City Campus, Nottingham
  - Queen Alexandra Hospital; Respiratory Centre, Portsmouth
  - Northern General Hospital, Sheffield
  - University Hospital of North Staffordshire; ILD Clinic, Stoke-on-Trent

REFERENCES:
- [Derived] Behr J, Nathan SD, Costabel U, Albera C, Wuyts WA, Glassberg MK, Haller H Jr, Alvaro G, Gilberg F, Samara K, Lancaster L. Efficacy and Safety of Pirfenidone in Advanced Versus Non-Advanced Idiopathic Pulmonary Fibrosis: Post-Hoc Analysis of Six Clinical Studies. Adv Ther. 2023 Sep;40(9):3937-3955. doi: 10.1007/s12325-023-02565-3. Epub 2023 Jun 30. PMID 37391667